CLINICAL TRIAL: NCT00527618
Title: A Randomized, Open-label, Crossover Trial of the Effect of Dosing of Daily HSV-2 Suppressive Therapy on HSV Reactivation and Plasma HIV-1 Levels Among HIV-1/ HSV-2 Co-infected Persons
Brief Title: Trial to Study the Effect of Dose of Herpes Simplex Virus-2 (HSV-2) Suppressive Therapy on HSV and HIV
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Jared Baeten, Principal Investigator, University of Washington
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 31203; GSK VAL111009 - VAL140 (Other Grant/Funding Number: GlaxoSmithKline)
Record Dates: First submitted 2007-09-07; First posted 2007-09-11 (Estimated); Results first posted 2012-07-31 (Estimated); Last update posted 2018-06-07 (Actual); Status verified 2018-05

CONDITIONS: Genital Herpes; HIV Infection
Keywords: Herpes Simplex Virus Type 2; Human Immunodeficiency Virus; Treatment Naive
MeSH Terms: conditions — Herpes Genitalis; HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Valacyclovir; Acyclovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard-dose acyclovir (Active Comparator): acyclovir 400 mg orally twice daily for 12 weeks.
  Interventions: Drug: acyclovir
- High-dose valacyclovir (Experimental): valacyclovir 1000 mg orally twice daily for 12 weeks.
  Interventions: Drug: valacyclovir

INTERVENTIONS:
Drug: valacyclovir — valacyclovir 1000 mg orally twice daily for 12 weeks.
  Other Names: Valtrex
  Arms: High-dose valacyclovir
Drug: acyclovir — acyclovir 400 mg orally twice daily for 12 weeks.
  Other Names: Zovirax
  Arms: Standard-dose acyclovir

SUMMARY:
To compare the effect of high-dose valacyclovir (1 gram orally twice daily) versus standard-dose acyclovir (400 mg orally twice daily) on the frequency of genital HSV reactivation and on plasma HIV-1 levels among HSV-2/HIV-1 co-infected individuals. The investigators hypothesize that high-dose valacyclovir will result in greater reduction in plasma HIV-1 and genital HSV reactivation.

DETAILED DESCRIPTION:
We propose to conduct a randomized, open-label, cross-over study of 38 individuals who are HIV-1 seropositive and HSV-2 seropositive. Both men and women will be recruited for the study. Participants must not be on antiretroviral therapy and must not be planning to initiate antiretroviral therapy during the anticipated study period. Participants will be randomized 1:1 to receive acyclovir 400 mg twice daily or valacyclovir 1000 mg twice daily. After 12 weeks on the initial treatment, each participant will be crossed over to the alternative treatment arm for 12 weeks. The treatment periods will be separated by a 2-week washout period. During the first four weeks of each treatment period (i.e. weeks 1-4 and weeks 15-18), participants will provide self-collected genital swabs daily for HSV DNA quantification. Each week during the entire study period plasma samples will be collected from participants for HIV-1 RNA quantification.

Open-label acyclovir and valacyclovir will be used for this trial, as the primary outcome measures (genital HSV and plasma HIV-1) are unlikely to be influenced by knowledge of treatment assignment. However, laboratory staff performing plasma HIV-1 and genital HSV measurements will not be aware of treatment assignment.

Optional Sub-Study A: Sub-study A will be offered to study participants. The purpose of sub-study A is to measure the effect of valacyclovir twice daily on plasma HIV-1 replication.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Documented HIV-1 seropositive
* Not on HIV-1 antiretroviral therapy nor planning to initiate antiretroviral therapy during the study period
* Detectable HIV-1 plasma viral load
* HSV-2 seropositive as determined by western blot
* Not intending to move out of the area for the duration of study participation
* Willing and able to provide independent written informed consent
* Willing and able to undergo clinical evaluations
* Willing and able to take study drug as directed
* Willing and able to adhere to follow-up schedule

Exclusion Criteria:

* Known history of adverse reaction to acyclovir, valacyclovir, or famciclovir
* Planned open label use of acyclovir, valacyclovir, or famciclovir
* History of evidence of CMV disease
* Known medical history of seizures
* Known renal insufficiency, defined as serum creatinine greater than 1.5 mg/dl
* AST or ALT greater than 3 times upper limit of normal
* Hematocrit less than 30 %
* Neutropenia, defined as absolute neutrophil count less than 1000
* Thrombocytopenia, defined as platelet count less than 75,000
* History of thrombotic microangiopathy
* For women, pregnancy as confirmed by a urine pregnancy test
* Any other condition which, in the opinion of the principal investigator, may compromise the ability to follow study procedures and complete the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2007-12; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jared Baeten, MD, PhD, Principal Investigator — University of Washington; Anna Wald, MD, MPH, Study Director — University of Washington
Locations (1):
- University of Washington Virology Research Clinic, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We recruited HIV-1/HSV-2 coinfected patients in Seattle, WA, between January 2008 and June 2010.
Pre-assignment Details: Of 49 persons screened, 15 were found to be ineligible for reasons including lack of HSV-2 infection (n=5), plans to initiate ART (n=3), undetectable plasma HIV-1 RNA (n=3), neutropenia (n=2), elevated hepatic transaminases (n=1), and incarceration (n=1). The remaining 34 participants were randomized.
Groups:
- Acyclovir Followed by Valacyclovir: Acyclovir 400 mg twice daily, followed by a two-week washout period, then valacyclovir 1000 mg twice daily
- Valacyclovir Followed by Acyclovir: Valacyclovir 1000 mg twice daily, followed by a two-week washout period, then acyclovir 400 mg twice daily
Period: Week 1-12 (First Intervention)
Arm/Group | Acyclovir Followed by Valacyclovir | Valacyclovir Followed by Acyclovir
Started | 16 (Acyclovir) | 18 (Valacyclovir; one participant was removed from the study due to urticaria after 2.5 weeks)
Completed | 13 (Acyclovir) | 16 (Valacyclovir)
Not Completed | 3 | 2
Not completed — Lost to Follow-up | 3 | 1
Not completed — Adverse Event | 0 | 1
Period: Week 13-14 (Washout)
Arm/Group | Acyclovir Followed by Valacyclovir | Valacyclovir Followed by Acyclovir
Started | 13 | 16
Completed | 12 | 16
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Period: Week 15-18 (Second Intervention)
Arm/Group | Acyclovir Followed by Valacyclovir | Valacyclovir Followed by Acyclovir
Started | 12 (Valacyclovir) | 16 (Acyclovir)
Completed | 12 (Valacyclovir) | 13 (Acyclovir)
Not Completed | 0 | 3
Not completed — Lost to Follow-up | 0 | 1
Not completed — Censored on initiation of HAART | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: This includes all 34 participants who were randomized. A subset of 28 participants were included in the analysis since only 28 participants contributed samples on both arms of the crossover study.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 34
Age, Continuous [Mean (Full Range); unit: Years] | 43 [24 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 28
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 23
  African-American | 9
  Other | 2
CD4 Count [Mean (Full Range); unit: cells/microliter] | 526 [73 to 1094]
Plasma HIV-1 RNA [Mean (Full Range); unit: log10 copies/mL] | 3.84 [1.17 to 6.93]

OUTCOME MEASURES:

1. Primary Outcome: The Quantity of HIV-1 RNA in Plasma While on 400 mg Twice Daily of Acyclovir Versus 1000 mg Twice Daily of Valacyclovir.
Description: Weekly measurements of plasma HIV-1 RNA on each drug were compared. The primary analysis was of the average difference in plasma HIV-1 RNA on valacyclovir and acyclovir as determined by a linear mixed model. The median of the average per-participant plasma HIV-1 RNA levels on valacyclovir and valacyclovir is also listed.
Time Frame: 26 weeks (12 weeks per drug intervention)
Population: Of the 34 participants who were randomized, 6 participants did not contribute to both arms of the study. The final analysis set therefore included 28 participants. 27 participants had plasma HIV-1 RNA levels available for analysis, since samples for one participant were persistently inhibited.
Measure: Median (Full Range); unit: log10 copies/mL
Groups:
- Acyclovir: Acyclovir, 400 mg orally twice daily (assigned to the acyclovir arm in either the first or second intervention periods)
- Valacyclovir: Valacyclovir, 1000 mg orally twice daily (assigned to the valacyclovir arm in either the first or second intervention periods)
Arm/Group | Acyclovir | Valacyclovir
Number analyzed (Participants) | 27 | 27
log10 copies/mL | 4.08 [1.17 to 5.33] | 3.68 [1.17 to 4.99]
Statistical Analysis 1: Comparison: Acyclovir vs Valacyclovir; We estimated that a sample size of 29 participants, with 4 weeks of weekly plasma HIV-1 RNA levels per treatment arm, would be required to detect a 0.25 log10 copies/ml difference in plasma HIV-1 RNA between the study arms with 80% power, at a two-sided type I error rate of 5%; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Adjusted for baseline plasma HIV-1 RNA; Slope = -0.27, 95% CI 2-sided [-0.41 to -0.14] — Acyclovir was coded as 0 and valacyclovir as 1. The beta-coefficient (slope) indicates the average difference in HIV-1 RNA on valacyclovir and acyclovir; a negative number indicates that plasma HIV-1 RNA was lower on valacyclovir than acyclovir

2. Primary Outcome: The Genital HSV Shedding Rate While on 400 mg Twice Daily of Acyclovir Versus 1000 mg Twice Daily of Valacyclovir.
Description: HSV DNA quantitated from daily self-collected genital swabs for the first four weeks of each drug intervention. The shedding rate was determined by the combined number of swabs with HSV detected divided by the combined number of swabs collected from participants, multiplied by 100.
Time Frame: The first four weeks of each intervention
Population: Of the 34 participants who were randomized, 6 participants did not contribute to both arms of the study. The final analysis set therefore included 28 participants.
Measure: Number; unit: percentage of swabs collected with HSV
Arm/Group | Acyclovir | Valacyclovir
Number analyzed (Participants) | 28 | 28
percentage of swabs collected with HSV | 8.2 | 7.8
Statistical Analysis 1: Comparison: Acyclovir vs Valacyclovir; We estimated that 26 participants would be required to detect a 50% reduction in genital HSV shedding with 80% power, at a two-sided type I error rate of 5%; Test type: Superiority or Other; p = 0.78, Random effects poission regression; Adjusted for age; Risk Ratio (RR) = 0.95, 95% CI 2-sided [0.66 to 1.37]

3. Secondary Outcome: The Effect of Valacyclovir 1 Gram Twice Daily Compared to Acyclovir 400 mg Twice Daily on the Percentage of Days With Genital Herpes Lesions.
Description: The percentage of days with genital herpes lesions was determined by the combined diary days in which genital lesions were recorded divided by the combined number of diary days for participants in the first four weeks of each drug intervention, multiplied by 100.
Time Frame: 26 weeks (12 weeks per drug intervention)
Population: as for outcome 2
Measure: Number; unit: percentage of days with genital lesions
Arm/Group | Acyclovir | Valacyclovir
Number analyzed (Participants) | 28 | 28
percentage of days with genital lesions | 4.0 | 1.0
Statistical Analysis 1: Comparison: Acyclovir vs Valacyclovir; Test type: Superiority or Other; p = 0.16, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: The Effect of Valacyclovir 1 g Twice Daily Compared With Acyclovir 400 mg Twice Daily on the Quantity of Genital HSV Detected During Shedding Episodes.
Description: HSV DNA was quantitated from daily self-collected genital swabs for the four weeks of each drug intervention. The quantity of genital HSV DNA present, when HSV DNA was detected, was compared.
Time Frame: The first four weeks of each intervention
Population: as for outcome 2
Measure: Median (Full Range); unit: log10 copies/mL
Arm/Group | Acyclovir | Valacyclovir
Number analyzed (Participants) | 28 | 28
log10 copies/mL | 3.0 [2.2 to 6.4] | 3.0 [2.2 to 6.8]
Statistical Analysis 1: Comparison: Acyclovir vs Valacyclovir; Test type: Superiority or Other; p = 0.67, Mixed Models Analysis

5. Secondary Outcome: Sub-Study: To Evaluate the Kinetics of Plasma HIV-1 Decline Over the First Three Days of High-dose Valacyclovir Administration.
Description: Plasma HIV-1 RNA was measured one day prior to, at initiation, and at 6, 24, 48, and 72 hours after initiating valacyclovir. Measurements at 24, 48, and 72 hours were used to determine the rate of HIV-1 RNA decline.
Time Frame: 72 hours
Population: In April 2010, we invited participants, including those who already completed the study, to participate in the substudy. Two participants had plasma HIV-1 RNA <40 copies/mL at the time of valacyclovir initiation and were excluded from analysis.
Measure: Mean (95% Confidence Interval); unit: log10 copies/mL/day
Groups:
- Valacyclovir: Valacyclovir, 1000 mg orally twice daily
Arm/Group | Valacyclovir
Number analyzed (Participants) | 10
log10 copies/mL/day | -0.20 [-0.38 to -0.19]

ADVERSE EVENTS:
Time Frame: 26 weeks
Description: Assessment of any adverse events was performed at each weekly clinic visit during the trial by a study investigator, including 12 weeks during acyclovir administration, 12 weeks during valacyclovir administration and 2 weeks during the washout period.
Arm/Group | Acyclovir | Valacyclovir
Serious Adverse Events (participants affected / at risk) | 1/32 | 0/30
Other Adverse Events (participants affected / at risk) | 4/32 | 3/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acyclovir (N=32) | Valacyclovir (N=30)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — One participant developed neutropenia on acyclovir: nadir ANC 570 cells/µL. This was thought to be related to concomitant interferon use. With cessation of interferon, the ANC normalized remaining normal with 12 weeks of high-dose valacyclovir.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acyclovir (N=32) | Valacyclovir (N=30)
Upper Resipiratory Tract Infection (Infections and infestations) | 4 (4) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 2 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3) | 1 (2)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Yeast vaginitis (Reproductive system and breast disorders) | 1 (3) | 2 (3)
Depression (Psychiatric disorders) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
Our findings are limited by the high loss to follow up, which is especially problematic in cross-over studies.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No